CLINICAL TRIAL: NCT06770296
Title: Pyrotinib at Different Doses in Combination With Trastuzumab and Paclitaxel Chemotherapy for First-Line Treatment of HER2-Positive Advanced Breast Cancer: A Multicenter, Randomized, Double-Cohort Study
Brief Title: The Dosing Regimen of Pyrotinib in HER2-positive Advanced First-line Breast Cancer: a Phase I Clinical Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The First People's Hospital of Xuzhou (Other); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); The Second People's Hospital of Changshu (Unknown); Shuyang County Traditional Chinese Medicine Hospital (Unknown); Affiliated Hospital of Nantong University (Other); Affiliated Hospital of Jiangsu University (Other); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Photine-01
Record Dates: First submitted 2024-12-19; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: HER2 positive; Pyrotinib
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyrotinib low dose group (Experimental): Pyrotinib: 320mg , peros(po) , once a day(qd) , every 3 weeks(q3w)
  Interventions: Drug: Pyrotinib low dose group
- Pyrotinib normal dose group (Active Comparator): Pyrotinib: 400mg , peros(po) , once a day(qd) , every 3 weeks(q3w)
  Interventions: Drug: Pyrotinib normal dose group

INTERVENTIONS:
Drug: Pyrotinib low dose group — Pyrotinib: 320mg, peros(po),once a day(qd) ,every 3 weeks(q3w) Trastuzumab: 8mg/Kg in the first cycle, 6mg/Kg in the subsequent cycle, intravenous(iv), every 3 weeks(q3w) Docetaxel: 75mg/m2，intravenous(iv), every 3 weeks(q3w)
  Arms: Pyrotinib low dose group
Drug: Pyrotinib normal dose group — Pyrotinib: 400mg, peros(po),once a day(qd) ,every 3 weeks(q3w) Trastuzumab: 8mg/Kg in the first cycle, 6mg/Kg in the subsequent cycle, intravenous(iv), every 3 weeks(q3w) Docetaxel: 75mg/m2，intravenous(iv), every 3 weeks(q3w)
  Arms: Pyrotinib normal dose group

SUMMARY:
Evaluate the safety and efficacy of Pyrotinib at different doses in combination with trastuzumab and paclitaxel chemotherapy for first-line treatment of HER2-positive advanced breast cancer.

DETAILED DESCRIPTION:
This study is planned to include 200 patients with HER2-positive advanced breast cancer meeting the admission criteria between 2024-11-01 and 2026-11-01. Statistical software will be used by the randomization officers for 1:1 allocation to pyrotinib 320mg in combination with trastuzumab and paclitaxel chemotherapy group and pyrotinib 400mg in combination with trastuzumab and paclitaxel chemotherapy group.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joins the study and signs the informed consent;
* Subject is an adult female or male ≥ 18 years old and ≤ 75 years old at the time of informed consent;
* HER2-positive advanced breast cancer confirmed by pathology:HER2-positive was defined as >10% of immunoreactive cells with an immunohistochemical (IHC) score of 3+ or HER2 gene amplification as a result of in situ hybridization (ISH). HER2 positivity should be verified by the pathology department of the research center;
* Recurrent or metastatic breast cancer; Patients with local recurrence had to be confirmed by the investigator as not amenable to curative resection;
* At least one measurable lesion or only bone metastases according to RECIST v1.1 criteria (including osteolytic lesions or mixed osteolytic/osteoblastic lesions);
* When randomized, Eastern Cooperative Oncology Group(ECGO) physical fitness status is 0 or 1 point;
* Vital organ function meets the following requirements (excluding the use of any blood components and cell growth factors during screening) : Absolute neutrophil (ANC) count ≥1.5×109/L; Platelet (PLT) ≥100×109/L; Hemoglobin (HB) ≥9g/dL; Total Bilirubin(TBIL) ≤ULN((Known patients with Gilbert's syndrome:Total Bilirubin(TBIL) ≤2×ULN);Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5×ULN(Patients with liver metastasis:ALT and AST≤5×ULN); Alkaline phosphatase (AKP) ≤ 2.5 times ULN; Blood Urea Nitrogen and Serum creatinine (Cr) ≤1.5×ULN;Left Ventricular Ejection Fractions(LVEF)≥50%;Corrected QT Interval(QTcF)<470msec.

Exclusion Criteria:

* The patient has received any systemic antitumor therapy at the stage of recurrence/metastasis, including any agents targeting EGFR or HER2, systemic chemotherapy, immunotherapy, and more than first-line endocrine therapy, as well as other antitumor therapies deemed by the investigators to be excluded;
* Tyrosine kinase inhibitor (TKI) preparations or macromolecular antibodies against HER have been used at any stage of breast cancer, except for trastuzumab in the (new) adjuvant stage;
* In the stage of breast cancer (new) adjuvant therapy, the time interval from the end of systemic therapy (except endocrine therapy) to the discovery of recurrence/metastasis is <12 months;
* Patients with active brain metastases with pial metastases confirmed by MRI or lumbar puncture (brain metastases requiring mannitol treatment or with symptoms);
* Grade≥ 3 peripheral neuropathy according to CTCAE4.0.3 criteria;
* Patients judged by the investigators to be unsuitable for systematic chemotherapy;
* Use of endocrine therapy drugs within 7 days prior to randomization;
* Patients with other malignancies within the previous 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma, or squamous cell carcinoma (patients with other malignancies occurring more than 5 years after randomization, such as those cured only by surgery, are allowed to be included);
* Had a major surgical procedure or significant trauma within 4 weeks prior to randomization, or was expected to undergo major surgery;
* Serious heart disease or discomfort, including but not limited to the following:

Previous history of heart failure or systolic dysfunction (LVEF<50%) High-risk or treatment-requiring angina pectoris or arrhythmias (e.g., second-degree type 2 atrioventricular block or third-degree atrioventricular block, ventricular tachycardia) Clinically significant valvular heart disease ECG showed transmural myocardial infarction Poor hypertension control (systolic blood pressure >150mmHg and/or diastolic blood pressure >100mmHg);

* Inability to swallow, chronic diarrhea, intestinal obstruction, or other factors affecting the administration and absorption of medications;
* Known allergic history of the drug components of this protocol;
* A history of immunodeficiency, including HIV infection, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
* Presence of third-space fluid accumulation that cannot be controlled by drainage or other methods (e.g., pleural fluid and ascites);
* Pregnant and lactating female subjects, or fertile subjects who were unwilling to use effective contraception throughout the trial period and within 3 months after the last study dose;
* Have a serious concomitant disease or other co-medical condition that interferes with planned treatment or any other condition that is not suitable for participation in this study, such as active hepatitis B, a lung infection requiring treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient is an adult female or male ≥ 18 years old and ≤ 75 years old at the time of informed consent.
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From the time of initiation of treatment in this study to the time of disease progression in the subjects,assessed up to 100 months.
  Objective Response Rate refers to the percentage of the total number of subjects in the analyzed data set who achieved the best response of CR or PR from the beginning of the study treatment to the time of the subject's disease progression group. Response Evaluation criteria in Solid Tumors (RECIST 1.1) was recommended to assess objective tumor response. Participants had to have measurable tumor lesions at baseline, and the response evaluation criteria were recommended as complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) according to RECIST 1.1 criteria.

OTHER OUTCOMES:
Progression Free Survival | From date of randomization until the date of first documented progression or death from any cause, whichever came first,assessed up to 100 months.
  Progression Free Survival refers to the time from the day of randomization until the first imaging assessment of disease progression (PD) or death from any cause. If subjects do not develop PD or die by the study deadline, or have received other antitumor therapy, the cut-off time will be based on the results of the last efficacy assessment before the deadline date or the start date of other antitumor therapy, whichever comes first.
Overall survival | From date of randomization until the date of first documented progression or death from any cause, whichever came first,assessed up to 100 months.
  Overall survival is defined as the time from the date of randomization to the date of death from any cause. For subjects who were still alive at the last follow-up, the OS was deleted based on the last follow-up time. For subjects who were lost to follow-up, the OS was calculated as the last confirmed survival time before the lost follow-up.
Duration of Response | From the first evaluation of CR, PR (whichever occurs first) to disease progression or death,whichever came first,assessed up to 100 months.
  Duration of Response refers to the time period from the first evaluation of CR, PR (whichever occurs first) to disease progression or death. RECIST 1.1 standard was used for evaluation.
Patient report outcome | Through study completion, an average of 1 year(From the date of enrollment to the clinical outcome from patients' report)
  The rating is evaluated by Functional Assessment of Cancer Therapy-Breast scale. It contains questions in five dimensions, with scores ranging from 0 to 4 for each question, with higher scores generally indicating a better quality of life
Incidence of Treatment-Emergent Adverse Events | From the beginning of the patient's use of pyrrotinib until the end of the safety follow-up period (28 days after the last dose).
  Adverse events include abnormal liver function, myelosuppression and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Yin, Ph.D, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No